CLINICAL TRIAL: NCT05726838
Title: A Belgian Registry to Evaluate the Real Life Treatment With Inclisiran on Top of Standard of Care Lipid-lowering Therapy in Patients With Atherosclerotic Cardiovascular Disease
Brief Title: The Belgian REAL (BE.REAL) Registry
Acronym: BE REAL
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839D1BE01
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: NIS; atherosclerotic cardiovascular disease; ASCVD; BE.REAL; BE REAL; inclisiran; Belgium
MeSH Terms: conditions — Atherosclerosis | interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Inclisiran: Patients prescribed inclisiran on top of standard of care lipid-lowering therapy
  Interventions: Other: Inclisiran

INTERVENTIONS:
Other: Inclisiran — There is no treatment allocation. Patients administered inclisiran by prescription will be enrolled. The patients will receive inclisiran therapy as per the approved label and Belgian reimbursement conditions.

SUMMARY:
This is an observational non-interventional study. The visit schedule is according to the routine clinical practice. Only data corresponding to study variables within the specified study period will be collected.

The study will recruit patients into one single cohort: Inclisiran in combination with other LLTs. The patients will receive Inclisiran therapy as per the approved label and Belgian reimbursement conditions.

DETAILED DESCRIPTION:
The study aims to assess the effectiveness, safety and adherence for Inclisiran in combination with lipid-lowering therapy (LLT) under conditions of routine clinical practice. The Inclisiran cohort will include patients receiving Inclisiran therapy as per the approved label independently of background Standard of Care (SoC) therapy. This study will include both primary data collection and secondary use of data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years or older.
2. Patients with Atherosclerotic Cardiovascular Disease (ASCVD) who are eligible for commercially available Leqvio, as defined by the reimbursement criteria:

   Patients with ASCVD documented by previous coronary heart disease (CHD), cerebrovascular disease or peripheral artery disease (PAD) and LDL-C ≥ 100mg/dL despite a treatment of min 6 weeks with max tolerated statin (unless intolerance or contra-indication) in combination with ezetimibe (unless intolerance or contra-indication).
3. Heterozygous Familial Hypercholesterolemia (HeFH) patients with documented ASCVD who are eligible for commercially available Leqvio.
4. Patients who provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who have received Inclisiran previously.
2. Patients participating in a clinical trial with investigational product.
3. Heterozygous Familial Hypercholesterolemia patients without established Atherosclerotic Cardiovascular Disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will consist of adult ASCVD patients and elevated levels of LDL-C with an initial prescription for Leqvio between 01-May-2022 and 31- Dec-2025, who provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean percent change in LDL-C from baseline | Baseline, up to 39 months
  Mean percent change in Low-Density Lipoprotein Cholesterol (LDL-C) from baseline will be collected
Mean absolute change in LDL-C from baseline | Baseline, up to 39 months
  Mean absolute change in Low-Density Lipoprotein Cholesterol (LDL-C) from baseline
Percentage of patients achieving the guideline-recommended LDL-C target at any time | Up to 39 months
  Percentage of patients achieving the guideline-recommended Low-Density Lipoprotein Cholesterol (LDL-C) target at any time will be collected

SECONDARY OUTCOMES:
Percentage of patients maintaining the guideline-recommended LDL-C target | Up to 39 months
  Percentage of patients maintaining the guideline-recommended LDL-C target (once achieved) for the duration of the study will be collected
Time- adjusted percentage change in LDL-C from baseline | Baseline, month 3, month 9, month 15, month 21, month 27, month 33, month 39
  time- adjusted percentage change in LDL-C from baseline to 3 months (2nd injection), 9 months (3rd injection), 15 months (4th injection), 21 months (5th injection), 27 months (6th injection), 33 months (7th injection) and 39 months (8th injection)
Change in LDL-C from baseline stratified on background therapy | Baseline, up to 39 months
  Change in LDL-C from baseline stratified on background therapy will be collected
Percentage of patients remaining on Inclisiran therapy at each injection visit | Up to 39 months
  Percentage of patients remaining on Inclisiran therapy at each injection visit will be collected
Percentage of patients with dose changes, switching, discontinuation | Up to 39 months
  Percentage of patients with dose changes, switching or discontinuation will be collected
Number of ASCVD-related events | Up to 39 months
  Number of atherosclerotic cardiovascular disease (ASCVD)-related events will be collected
Number of possibly related adverse events | Up to 39 months
  Number of possibly related adverse events will be collected
Number of injection site reactions | Up to 39 months
  Number of injection site reactions will be collected
Number of patients with changes in Lp(a) levels for Inclisiran-treated patients | Up to 39 months
  Number of patients with changes in Lipoprotein (a) levels for Inclisiran-treated patients will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Belgium (15):
  - Novartis Investigative Site, Turnhout, Antwerpen
  - Novartis Investigative Site, Yvoir, Namur
  - Novartis Investigative Site, Kortrijk, West-Vlaanderen
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Anderlecht
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Haine-Saint-Paul
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Mechelen

IPD SHARING:
Plan to Share IPD: No